CLINICAL TRIAL: NCT07121530
Title: Role Of Human Papilloma Virus In Male Infertility In Qena Government - Upper Egypt
Brief Title: Human Papilloma Virus In Male Infertility
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Abderlraheem Abdellatif, Resident at Dermatology , venereology and andrology, Faculty of medicine, South Valley University
Other Study IDs: SVU-MED-DVA021-1-23-8-706
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2023-08

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile Males Group: About 30 infertile males with genital wart
  Interventions: Procedure: HPV infection in infertile males
- Control Group: About 20 healthy males
  Interventions: Procedure: HPV infection in infertile males

INTERVENTIONS:
Procedure: HPV infection in infertile males — To investigate the status of HPV infection in infertile males in Qena government, and to Analyse the effects of HPV infection on semen parameters.
  Other Names: infertile males

SUMMARY:
Infertility is a major health problem worldwide and is estimated to affect 8-12% of couples in the reproductive age group.

Infertility affects both men and women. Male causes for infertility are found in 50% of these couples.

HPV may infect the semen ,allowing it to affect male fertility in a variety of ways.

DETAILED DESCRIPTION:
WHO defines infertility as the inability to conceive after at least 12 months of regular, unprotected sexual intercourse.

Reduced male fertility can be the result of congenital and acquired urogenital abnormalities, infections of the male accessory glands, increased scrotal temperature (varicocele), endocrine disturbances, genetic abnormalities and immunological factors ,

In 40-60% of cases the only abnormality is the semen analysis and there is no relevant history or abnormality on physical examination and endocrine laboratory testing (idiopathic male infertility).

Semen analysis reveals a decreased number of spermatozoa (oligozoospermia), decreased motility (asthenozoospermia) and many abnormal forms on morphological examination (teratozoospermia). Usually, these abnormalities come together and are described as the OAT-syndrome (oligo-astheno-teratozoospermia).

Human papillomavirus (HPV) is one of the most common sexually transmitted viruses, and males and females from different regions are generally susceptible.

More than 120 HPV genotypes are known to distribute in the skin and mucous membranes, including the pubic area, oral cavity and perianal region, and can be transmitted through skin contact or any other surface contact related to the genital area.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 year of unprotected sexual intercourse without conception.
* Patients with genital warts

Exclusion Criteria:

* Hypergonadotropic/hypogonadotropic hypogonadism
* Azoospermia
* chromosome abnormalities
* undescended testis
* mumps orchitis

Ages: 23 Years to 53 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted (30)infertile males with genital wart ,control (20) attending the Dermatology, Venereology& Andrology clinic in Qena University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Investigation of Human Papilloma Virus infection in infertile males | 2 Days
  Investigation of Human Papilloma Virus (HPV) infection in infertile males as : all participants in the study made semen analysis and the semen were collected by masturbation after 5-7 days of abstinence. Semen parameters (semen volume, sperm concentration, progressive motility (PR) and rate of normal sperm morphology) were analyzed in a thermostat console after semen liquefaction. then Seminal Detection of HPV antibodies in infertile male by HPV ELISA Kit and also to see its effects on semen parameters in Qena government.

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Professor, Study Chair — Dermatology, Venereology and Andrology. Faculty of Medicine,South ValleyUniversity
Locations (1):
- Qina University hospital, South Valley University Hospital, Qina, Egypt